CLINICAL TRIAL: NCT04847414
Title: Novel Classification of Adult-onset Diabetes and Its Association With Common Microvascular Complications in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Faysal Elrawy Refaie, assistant lecturer, The principal investigator, Sohag University
Other Study IDs: Soh-Med-21-04-16
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective group: all needed data will be collected from patients in this group through performing full medical examination and doing all necessary investigations for them
  Interventions: Diagnostic Test: HbA1C, other investigations
- retrospective group: all needed data will be collected from medical records either electronic or paper based from different diabetes clinics in upper Egypt

INTERVENTIONS:
Diagnostic Test: HbA1C, other investigations — we will do some necessary investigations for prospective group
  Groups: prospective group

SUMMARY:
Aim of our work:

First aim: Classify patients with adult-onset diabetes according to the novel classification into new subgroups, depending on multiple variables related clinically to those patients.

Second aim: To identify the association between the new classification subgroups and the presence of common microvascular complications (retinopathy, nephropathy, and neuropathy), which can help in the early prediction of these complications and their early management.

DETAILED DESCRIPTION:
We will conduct an observational cross-sectional study and cluster analysis for patients from different Diabetes clinics and tertiary centres located in different governorates in Upper Egypt. Our participants in this study will be divided into two groups:

1. The first group will be as a prospective group, All necessary examinations and investigations will be performed for every patient of this group during their clinic visit at the time of registration to this study.
2. The second group will be the retrospective group. Data for those patients will be collected from electronic records and/or paper records in collaboration with different diabetes centres and clinics scattered in Upper Egypt governorates. We will collect clinical and lab data as much as we can. All available data for this group at end of this study will be used in the clustering of this group.

Then we will use the above data from both groups to classify diabetic patients to the new clusters and to find the association between those clusters and the incidence of microvascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult-onset DM type 2 diagnosed patients according to current ADA recommendations, aged <18 years old and within 3 years from the time of diagnosis.

Exclusion Criteria:

* 1- Patients diagnosed with Gestational DM or rare types of diabetes like monogenic diabetes types, such as maturity-onset diabetes of the young (MODY), diabetes secondary to steroid use, cystic fibrosis, hemochromatosis, and pancreatic diabetes according to ADA criteria.

  2- Patients diagnosed with non-diabetic kidney diseases, such as chronic glomerulonephritis, vasculitis, polycystic kidney disease, and renal cancer or patients with a transplanted kidney were excluded from the analysis for diabetic kidney disease.

  3- Patients diagnosed with retinopathy due to non-diabetic causes or diagnosed with neuropathy due to non-diabetic causes will be excluded from the analysis for diabetic retinopathy and neuropathy, respectively.

Ages: 18 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients diagnosed with diabetes within 3 years in Upper Egypt
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2023-04-24 (Estimated); Study Completion 2023-04-24 (Estimated)

PRIMARY OUTCOMES:
change in HbA1C | 3 months
  percent %
change in BMI | 3 months
  kg/m2

SECONDARY OUTCOMES:
HOMA-IR | 6 months
  calculated by HOMA calculator presented by Oxford University

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
sharing final results only